CLINICAL TRIAL: NCT04353154
Title: Development and Evaluation of Applying a Point-of-Care COVID-19 Test Strategy to Triage Patients Presenting with Acute Coronary Syndromes, Respiratory or Hemodynamic Instability and Out of Hospital Cardiac Arrests
Brief Title: The RAPID COVID-19 TRIAGE Algorithm
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 20200228-01H
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Spartan Cube Point-of Care Covid-19 test — Throat and nasal swab for COVID-19 point-of-care test.

SUMMARY:
This study is being conducted to study the use and application of a point-of-care (POC) Covid-19 test developed by Spartan BioSciences and recently approved for clinical use by Health Canada. Phase I of this study will determine the best route for the swabs (nasal, throat, or both), and to determine if this POC test results are comparable to the standard core-lab test results.

DETAILED DESCRIPTION:
Currently, testing for COVID-19 is carried out with swabs and blood tests that are sent to hospital laboratories for analysis. With the current technology, the turnaround time for test results may take any where from 8 hours up to several days for confirmation of whether you have COVID-19. This delay in diagnosis may delay care, prevent other testing modalities, consume isolation beds and deplete the valuable personal protective equipment (PPE) needed while providing treatment for patients with COVID-19.

Using a new, Health Canada approved technology, we can conduct the virus genetic testing at the bedside with a nostril and throat swab, with results in under 45 minutes. This new "point-of-care (POC)" technology, if proven accurate, may help future patients receive faster and more definitive treatment. At the same time, it might help health care teams to preserve resources and optimize care for patients (example: triage use of intensive care or isolation unit beds, determine need for PPE, get quarantined staff back to front line to help with care if they are non-carriers).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 yo referred to the cardiology, internal medicine, ICU, CICU, CSICU or RACE teams who have tested positive for COVID-19.

Exclusion Criteria:

* Patients in whom conventional COVID-19 testing would not have otherwise been instituted or in whom immediate test results would not alter short-term treatment, Patients with pre-existing wishes for DNR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is admitted patients who have had a positive core-lab virology test for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 1 month
  For the analysis, this will be based on a comparison of the identified patients in the core lab with the POC testing with the following data to arrive at an early sensitivity:
  Sensitivity = True Positive/ (True positive/True positive + False Negative)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No